CLINICAL TRIAL: NCT03190980
Title: Efficacy and Safety of Oral Glucose in Pain Alleviation Among Healthy Term Neonates
Brief Title: Oral Glucose in Pain Alleviation Among Term Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Amal Naous, Pediatrician, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 1722017
Record Dates: First submitted 2017-06-13; First posted 2017-06-19 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 5% glucose (Experimental): neonates will receive 2 ml of 5% glucose before heel prick
  Interventions: Other: 5% glucose
- 30% glucose (Experimental): neonates will receive 2 ml of 30% glucose before heel prick
  Interventions: Other: 30% glucose
- Placebo (Placebo Comparator): neonates will receive 2 ml of sterile water before heel prick
  Interventions: Other: Placebo

INTERVENTIONS:
Other: 5% glucose — Neonates will receive 5% glucose, then heel prick wil be performed during which pain will be assessed
  Arms: 5% glucose
Other: 30% glucose — Neonates will receive 30% glucose, then heel prick wil be performed during which pain will be assessed
  Arms: 30% glucose
Other: Placebo — Neonates will receive sterile water, then heel prick wil be performed during which pain will be assessed
  Arms: Placebo

SUMMARY:
Background: It was long believed that newborns could not experience pain. As it is now documented that newborns have all the necessary systems to perceive pain, pain management can no longer be ignored.

Pharmacologic agents are not recommended in neonates for pain relief in minor procedures and still there is debate regarding the efficacy of oral glucose, in different strengths, on alleviation of pain among neonates.

Aim: The objective of this study is to assess the efficacy and safety oral administration of glucose, in different concentrations, on pain relief in full term neonates undergoing heel prick test.

Methods: The investigators will conduct a prospective, randomized, double blind placebo controlled trial to investigate the effect of glucose solution on alleviating the pain of heel prick test in 244 healthy full term newborns who will be randomly allocated to one of three groups: First group will receive 5% glucose, second group will receive 30% glucose and third group will receive sterile water as a placebo, 2 minutes prior to the procedure.

Specially trained nurses will take turns to carry out blood sampling. Neonatal pain will be assessed by the Neonatal Infant Pain (NIPS) as well as by duration of crying, changes in heart rate, respiratory rate and oxygen saturation.

DETAILED DESCRIPTION:
The investigators will conduct a prospective, randomized, double blind, placebo controlled study of healthy full term newborns delivered by normal vaginal delivery, undergoing heel prick test. They will be randomized to receive either 5% glucose, 30% glucose or sterile water as a placebo, 2 minutes prior to the procedure. The investigators will study the efficacy and safety of oral glucose, in different strengths, compared to placebo (sterile water) in pain alleviation.

All parents will receive an explanation of the study before participation, and informed written consent will be signed by the parents for voluntary participation

ELIGIBILITY:
Inclusion Criteria:

* Estimated gestational age: 37 weeks-42 weeks
* Birth weight: 2500 grams- 4000 grams
* Mode of delivery: normal vaginal delivery
* Age: birth to 72 hours of life
* Apgar scores of at least 7 at 1 and 5 minutes
* Heart rate between 100 and 160 per minutes
* Blood O2 saturation ≥ 95%
* No known congenital anomalies

Exclusion Criteria:

* They have history of birth trauma
* They are admitted to neonatal intensive care unit (NICU)
* They need respiratory support
* Their mothers are receiving sedatives or opioids during vaginal delivery

Ages: 24 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 244 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Pain score | 2 minutes during the procedure
  Pain responses will be evaluated using the Neonatal Infant Pain Scale NIPS

SECONDARY OUTCOMES:
Occurance of adverse events | 5 minutes after the procedure
  local bruising or haematoma or hyperglycemia

CONTACTS AND LOCATIONS:
Locations (1):
- Makassed General Hospital, Beirut, Lebanon